CLINICAL TRIAL: NCT01725789
Title: A Randomized Patient -Blind Controlled Phase III Study to Compare the Efficacy and Safety of Intravenous Ferric Carboxymaltose (Ferinject®) With Placebo in Patients With Acute Isovolemic Anemia After Gastrectomy
Brief Title: Ferinject® Assessment In GastRectomy Patients With Acute Isovolemic Anemia (FAIRY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Woo Kim, Head of Department of Gastric Cancer Research, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCCCTS-12-644
Record Dates: First submitted 2012-11-03; First posted 2012-11-14 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Anemia
Keywords: Acute isovolemic anemia after gastrectomy for gastric cancer
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferinject® Group (Experimental): Ferinject®to be administered as IV drip infusion or undiluted bolus injection to consented patients with 7g/dl≤Hb<10g/dl at 5 - 7 days after gastrectomy for gastric cancer.
  Interventions: Drug: Ferinject®
- Placebo Group (Placebo Comparator): Placebo(0.9% Normal Saline) to be administered as IV drip infusion or bolus injection to consented patients with 7g/dl≤Hb<10g/dl at 5 - 7 days after gastrectomy for gastric cancer.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Ferinject® — Ferinject®to be administered as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg single administration) for body weight ≥50 Kg or 6 minutes (for 500mg single administration) for body weight <50Kg .
  Note, Ferinject® should be administered to a maximum of 20mg iron/kg. Therefore in patients with a body weight <50kg, administration of Ferinject® should be limited to 500mg at baseline . All patients with a serum ferritin value <15ng/mL and Hb<10g/dl at week 3 visit that a second dose (of 500mg iron or equivalent placebo) will be given.(Study group: Ferinject®500mg, Control Group:Placebo)
  Other Names: Ferric carboxymaltose
  Arms: Ferinject® Group
Drug: normal saline — Placebo will be in the form of normal saline administered over same time period as equivalent Ferinject® administration. IV drip infusion or undiluted bolus injection with a minimum administration time of 15 minutes (200mL as infusion or 20mL as bolus injection) for body weight ≥50 Kg or 6 minutes (100mL normal as infusion or 10mL as bolus injection) for body weight <50 Kg.
  Arms: Placebo Group

SUMMARY:
This study is designed to evaluate the efficacy of Ferinject® in improving acute isovolemic anemia after gastrectomy for gastric cancer in terms of Quality of life(QOL )and objective measures (Hb and iron parameters).

Furthermore, the tolerability and safety of Ferinject® treatment will be evaluated.

DETAILED DESCRIPTION:
Randomized patient-blind placebo controlled study. Hb level of 10 g/dl will be used as a cut-off value for our study based on the guidelines published by American Society of Clinical Oncology and the American Society of Hematology for the treatment of cancer-related anemia, recommending Hb<10 g/dl as a treatment threshold.

Ferinject® to be administered based on Hb and body weight per approved summary of product characteristics (SmPC).

5 - 7 days after gastrectomy for gastric cancer, consented patients with 7g/dl≤Hb<10g/dl will be administered Ferinject® or placebo (normal saline) based on the results of randomization.

• Study Group Ferinject®to be administered as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg single administration) for body weight ≥50 Kg or 6 minutes (for 500mg single administration) for body weight <50Kg .

Note, Ferinject® should be administered to a maximum of 20mg iron/kg. Therefore in patients with a body weight <50kg, administration of Ferinject® should be limited to 500mg at baseline . All patients with a serum ferritin value <15ng/mL at week 4 visit that a second dose (of 500mg iron or equivalent placebo) will be given.(Study group: Ferinject®500mg, Control Group:Placebo)

• Control Group Placebo will be in the form of normal saline administered over same time period as equivalent Ferinject® administration. IV drip infusion or undiluted bolus injection with a minimum administration time of 15 minutes (200mL as infusion or 20mL as bolus injection) for body weight ≥50 Kg or 6 minutes (100mL normal as infusion or 10mL as bolus injection) for body weight <50 Kg.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years old
* 7g/dl ≤ Hb < 10g/dl at 5 - 7 days after gastrectomy for gastric cancer
* signed written informed consent

Exclusion Criteria:

* a concurrent medical condition(s) that would prevent compliance or participation or jeopardize the health of the patient
* hypersensitivity to any component of the formulation
* active severe infection/inflammation
* History of transfusion, erythropoietin, > 500 mg intravenous iron administration within 4 weeks prior to screening.
* History of acquired iron overload.
* Pregnancy or lactation.
* Decreased renal function (defined as creatinine clearance < 50 mL/min calculated by Cockcroft-Gault)
* Chronic liver disease or increase of liver enzymes (ALT, AST) > 3 times the upper limit of normal range.
* Participation in any other interventional study within 1 month prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
• Number of responders | 12 weeks post baseline
  • Number of responders (Hb increase ≥2 g/dL with respect to the baseline Hb value and/or Hb ≥11g/dL ) by 12 weeks (independent of alternative anaemia management including transfusion or ESA use). Note, if patient requires an ESA or blood transfusion by week 12 will be considered a non-responder.

SECONDARY OUTCOMES:
• Percentage of patients with Hb ≥10, 11 and 12 g/dL | 3weeks , 12 weeks post baseline
  • Percentage of patients with Hb ≥10, 11 and 12 g/dL at 3 and 12 weeks (independent of alternative anaemia management including transfusion or ESA use)
• Percentage of patients requiring alternative anaemia management therapy | 12 weeks post baseline
  • Percentage of patients requiring alternative anaemia management therapy
• Self-reported patient assessment of EORTC QLQ C-30 and Sto-22 | 3weeks, 12weeks post baseline
  • Self-reported patient assessment of EORTC QLQ C-30 and Sto-22 at 3 weeks and 12 weeks
• Evolution of Hb, ferritin and TSAT | 12 weeks post baseline
  • Evolution of Hb, ferritin and TSAT over the study duration (12weeks) independent of alternative anaemia management including transfusion or ESA use
• adverse events: type, nature, incidence and outcome | up to 3 weeks post baseline
  • adverse events: type, nature, incidence and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Young Woo Kim, PhD, Principal Investigator — National Cancer Center, Rep. of Korea
Locations (6):
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun, Chollanam Do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Kyungpook national university hospital, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University, Seoul

REFERENCES:
- [Derived] Kim YW, Bae JM, Park YK, Yang HK, Yu W, Yook JH, Noh SH, Han M, Ryu KW, Sohn TS, Lee HJ, Kwon OK, Ryu SY, Lee JH, Kim S, Yoon HM, Eom BW, Choi MG, Kim BS, Jeong O, Suh YS, Yoo MW, Lee IS, Jung MR, An JY, Kim HI, Kim Y, Yang H, Nam BH; FAIRY Study Group. Effect of Intravenous Ferric Carboxymaltose on Hemoglobin Response Among Patients With Acute Isovolemic Anemia Following Gastrectomy: The FAIRY Randomized Clinical Trial. JAMA. 2017 May 23;317(20):2097-2104. doi: 10.1001/jama.2017.5703. PMID 28535237
- [Derived] Reim D, Kim YW, Nam BH, Kim MJ, Yook JH, Park YK, Roh SH, Yu WS, Bae JM. FAIRY: a randomized controlled patient-blind phase III study to compare the efficacy and safety of intravenous ferric carboxymaltose (Ferinject(R)) to placebo in patients with acute isovolemic anemia after gastrectomy - study protocol for a randomized controlled trial. Trials. 2014 Apr 5;15:111. doi: 10.1186/1745-6215-15-111. PMID 24708660